CLINICAL TRIAL: NCT00184938
Title: Opioid Induced Acute Preconditioning
Brief Title: Opioid Receptors Influence Ischemia-Reperfusion Injury
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: OPIRI
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Ischemia-Reperfusion Injury
Keywords: opioids; ischemic preconditioning; morphine
MeSH Terms: conditions — Reperfusion Injury | interventions — Morphine; Naloxone

INTERVENTIONS:
Drug: morphine
Drug: naloxone
Drug: Technetium-TC99m-labeled Annexin A5
Procedure: forearm ischemic exercise
Procedure: ten minute forearm ischemia

SUMMARY:
The most powerful protective mechanism against ischemia-reperfusion injury other than rapid reperfusion is ischemic preconditioning. Ischemic preconditioning is defined as the development of tolerance to ischemia-reperfusion injury by a previous short bout of ischemia resulting in a marked reduction in infarct size. This mechanism can be mimicked by several pharmacological substances such as adenosine and morphine.

We, the researchers at Radboud University Nijmegen Medical Centre, have recently developed a method in which we can detect ischemia-reperfusion injury in the human forearm by using Annexin A5 scintigraphy (Rongen et al). With this method we will determine whether opioid receptors are involved in ischemic preconditioning. We expect to find that morphine can mimic ischemic preconditioning and that acute ischemic preconditioning can be blocked with the opioid receptor antagonist naloxon. This study will increase our knowledge about the mechanism of ischemic preconditioning and may also provide leads to exploit this endogenous protective mechanism in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Exposition to radiation due to imaging techniques in the previous five years

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-01

PRIMARY OUTCOMES:
Percentual difference in Annexin A5 targetting between the experimental and control arm 1 and 4 hours after intravenous injection

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, Phd, Principal Investigator — Radboud University Nijmegen Medical Centre / Department of Pharmacology and Toxicology
Locations (1):
- Radboud University Nijmegen Medical Centre / Department of Pharmacology and Toxicology, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546